CLINICAL TRIAL: NCT03331588
Title: Comparison Study of Post-operative Pain and Quality of Life Between Subxiphoid and Intercostal Vedio-assisted Thoracic Surgery for Radical Lung Cancer Resection
Brief Title: Comparison of Post-operative Pain and Quality of Life Between Subxiphoid and Intercostal VATS for Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Lei Jiang, associate chief physician, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: leijiang
Record Dates: First submitted 2017-11-01; First posted 2017-11-06 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Lung Neoplasms; Thoracic Surgery; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Carcinoma, Bronchogenic; Thoracic Neoplasm
Keywords: Lung cancer; Pain; Quality of life
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Carcinoma, Bronchogenic; Thoracic Neoplasms; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider
Masking Description: In the operating room a dressing will be placed so that it covers the entire hemithorax whereby the incision is hidden. This is done identically regardless of surgical technique. This dressing is left in place until discharge. If changing of the dressing is needed, either the project-nurse or a nurse for another team will assist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subxiphoid uniportal VATS (Active Comparator): Standard Subxiphoid single-port video assisted thoracic surgery, no use of rib-spreader.
  Interventions: Procedure: Subxiphoid uniportal VATS
- Intercostal uniportal VATS (Active Comparator): Standard Intercostal single-port video assisted thoracic surgery, no use of rib-spreader.
  Interventions: Procedure: Intercostal uniportal VATS

INTERVENTIONS:
Procedure: Subxiphoid uniportal VATS — Patients were placed in a supine position, and the operating table was manipulated as needed to elevate the appropriate side of the body for surgery. The surgical procedures followed principles of pulmonary resections
  Arms: Subxiphoid uniportal VATS
Procedure: Intercostal uniportal VATS — The surgical procedures followed principles of pulmonary resections
  Arms: Intercostal uniportal VATS

SUMMARY:
One-thirds of patients underwent video-assisted thorascopic surgery (VATS) still have severe pain.Uniportal lobectomy or segmentectomies emerged as a promising and exciting approach for minimally invasive thoracic surgery. However, nearly all reported uniportal VATS lobectomies have been performed via the intercostal route, and chest wall trauma has still occurred. Here,the investigators undertook novel uniportal VATS technique involving a subxiphoid route for pulmonary lobectomies or segmentectomies.We would like to evaluate the post-operative pain and quality of life between Subxiphoid and Intercostal VATS for Lung Cancer.

DETAILED DESCRIPTION:
Is subxiphoid route VATS surgery better than Intercostal VATS surgery for lung cancer?

Video assisted thoracoscopic surgery for lung cancer (VATS) is less traumatic than traditional open surgery for lung cancer. A novel uniportal VATS technique involving a subxiphoid route for thoracic surgery has been occured. It is reported that subxiphoid route VATS surgery is better than Intercostal VATS surgery in post-operative pain and quality of life, but this has never been documented in a randomized trial. Some surgeons hesitate to use subxiphoid VATS because it is technically more demanding, others question if the two methods are oncologically equal. Regardless, VATS has been implemented as a routine method for lung cancer surgery several places around the world, while Shanghai pulmonary Hospital is one of the best to perform subxiphoid VATS. The investigators have launched the first randomized controlled trial in the world comparing the two surgical methods to investigate any differences in length of hospitalization, postoperative pain, life quality within the first year.

The investigators include patients with stage I lung cancer, and randomize between subxiphoid VATS and Intercostal VATS in a design where both the patient and doctors doing general rounds in the ward are blinded until discharge because the dressing on the surgical wound is identical, regardless of the surgical method. The surgeon cannot influence clinical decisions including time to discharge, which is decided by other specialist surgeons. Pain evaluation is performed 1 time daily and followed 6 months using the VAS-score, life quality is evaluated continuously during the first 6 months using SF-MPQ-2 questionnaires.

200 patients will be asked to participate in each study at shanghai pulmonary Hospital,china in collaboration with surgeons from department of thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for surgery for lunge cancer.

Elective surgery (surgery planed > 2 days).

Accepts randomization.

Age 18 or above.

Exclusion Criteria:

* Previous thoracic surgery.

Any type of chronic pain, requiring daily use of analgetics.

pregnant.

Breast feeding.

contraindications to NSAID.

Chemo- and/or radiotherapy in connection to present admission.

Major surgery planned in connection to this admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 6 months
  visual analogue score (VAS-score) is to asses the development of acute and chronic pain after VATS surgery. 11 point numeric rating scale of 0 represented "no pain"and a score of 10 represented "worst pain ".

SECONDARY OUTCOMES:
Quality of life | 6 months
  SF-MPQ-2 questionnaire is used.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gonzalez-Rivas D, Yang Y, Lei J, Hernandez L, Jiang G. Subxiphoid uniportal video-assisted thoracoscopic middle lobectomy and anterior anatomic segmentectomy (S3). J Thorac Dis. 2016 Mar;8(3):540-3. doi: 10.21037/jtd.2016.02.63. PMID 27076952
- [Background] Hernandez-Arenas LA, Lin L, Yang Y, Liu M, Guido W, Gonzalez-Rivas D, Jiang G, Jiang L. Initial experience in uniportal subxiphoid video-assisted thoracoscopic surgery for major lung resections. Eur J Cardiothorac Surg. 2016 Dec;50(6):1060-1066. doi: 10.1093/ejcts/ezw189. Epub 2016 Jul 11. PMID 27401700
- [Background] Song N, Zhao DP, Jiang L, Bao Y, Jiang GN, Zhu YM, Ding JA. Subxiphoid uniportal video-assisted thoracoscopic surgery (VATS) for lobectomy: a report of 105 cases. J Thorac Dis. 2016 Mar;8(Suppl 3):S251-7. doi: 10.3978/j.issn.2072-1439.2016.02.32. PMID 27014471
- [Derived] Chen Z, Jiang L, Zheng H, Zhang W, Lv X, Abdellateef A. Early postoperative pain after subxiphoid uniportal thoracoscopic major lung resection: a prospective, single- blinded, randomized controlled trial. Interact Cardiovasc Thorac Surg. 2022 Jun 15;35(1):ivac133. doi: 10.1093/icvts/ivac133. PMID 35579360